CLINICAL TRIAL: NCT03405038
Title: Prone Position Impact in Patients With Acute Respiratory Distress Syndrome on the Incidence of Central Venous Catheter Colonizations in Reanimation
Brief Title: Prone Position Impact in ARDS Patients on the Incidence of Central Venous Catheter Colonization
Acronym: ILCDV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-02-CHRMT
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2018-01

CONDITIONS: ARDS, Human; Catheter Infection
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Catheter colonization, catheter-associated infection and catheter-associated bacteremia are a major challenge for resuscitation unit. This study wishes to explore the impact of the central venous catheter colonization on the ARDS patient with and without prone position.

DETAILED DESCRIPTION:
Catheter-associated infection prevention is achieved by identification of the population at risk. Patients receiving prone position Under acute respiratory distress syndrome appear to be particularly vulnerable. This retrospective study is designed to compare the risk of catheter colonization that could be induced or worsened by prone position. Knowing that, prone position is increased into the care acute respiratory distress syndrome since few years. Unfortunately, no study has examined the prone position impact on catheter-association infection in these population.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patient in the reanimation unit of the CHR Metz-Thionville or the CHRU Nancy between january 2014 and december 2015
* Patient with an acute respiratory distress syndrome, moderate or severe
* With a central venous catheter
* With or without prone position during the stay

Exclusion Criteria:

* Minor patient
* Absence of information on central venous catheter bacteriology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ARDS patients with a central venous catheter placed or not into prone position
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Impact of the prone position | Day 1
  Incidence rate of the bacterial colonization at least one catheter during the stay in resuscitation unit

SECONDARY OUTCOMES:
Infection associated factors | Day 1
  multivariate analysis of risks factor for the catheter colonization ((age, sex, comorbidity, weight, length of stay)

CONTACTS AND LOCATIONS:
Locations (1):
- CHR Metz Thionville, Metz, France